CLINICAL TRIAL: NCT02161471
Title: Haemodynamics and Function of the Atria in Patients With Congenital Heart Defects - Pilot Study by Cardiovascular Magnetic Resonance
Brief Title: Haemodynamics and Function of the Atria in Congenital Heart Disease by Cardiovascular Magnetic Resonance
Status: Completed | Type: Observational
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: Atrial function in CHD by CMR
Record Dates: First submitted 2014-06-10; First posted 2014-06-11 (Estimated); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Coarctation of the Aorta; Tetralogy of Fallot; Transposition of the Great Arteries
Keywords: Atria, Heart; Function, Atrial; Heart Defects, Congenital; Cardiovascular Abnormalities; Congenital Abnormalities; Tetralogy, Fallot; Transposition of Great Arteries; Coarctation of the Aorta
MeSH Terms: conditions — Aortic Coarctation; Tetralogy of Fallot; Transposition of Great Vessels; Heart Defects, Congenital; Cardiovascular Abnormalities; Congenital Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Tetralogy of Fallot: Patients after repair of tetralogy of Fallot
- Normal: Normal controls

SUMMARY:
The purpose of this study is to determine whether patients with repaired congenital heart disease show differences in size or function of their heart atria compared to normal controls and depending on the nature of their heart disease.

DETAILED DESCRIPTION:
Atrial function is important for good ventricular filling and function. In patients with impaired cardiac function, atrial contraction is even more important. So far, the size and function of the atria have been assessed two-dimensionally by angiography and by echocardiography. However, these do not allow exact characterization of the volumetric changes of the atria during the cardiac cycle. Recently, cardiac magnetic resonance (CMR) has been used to assess size and function of the left atrium in adults. Little data are available about function and volume of the atria in children and the role of the atria in congenital heart disease (CHD).

The study will recruit patients with CHD (n=40) and normal controls (n=10). The patient group will be composed by patients suffering from the following conditions: coarctation of the aorta (n=10), tetralogy of Fallot (n=10), transposition of the great arteries after atrial switch (Senning procedure) (n=10), transposition of the great arteries after arterial switch operation (n=10).

The study consists of measurements of sizes and function of the right and the left atrium, respectively, by examining three-dimensional volume changes across the heart cycle, and of phase contrast measurements of blood flow across the valves of the heart.

ELIGIBILITY:
Inclusion Criteria:

* Ability to perform repetitive breath holds of 10-15 seconds each
* Written informed consent of the patients or their legal guardians

Exclusion Criteria:

* Patients requiring general anaesthesia
* Residual cardiac findings which might potentially influence the size and function of the atria

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants for the study will be recruited among patients, children and adults, with CHD (groups 1-4) undergoing cardiac magnetic resonance examination for clinical reasons.
  1. Patients after repair of coarctation of the aorta
  2. Patients after repair of tetralogy of Fallot
  3. Patients with transposition of the great arteries after atrial switch (Senning procedure)
  4. Patients with transposition of the great arteries after arterial switch operation
  5. Children without cardiovascular anomalies undergoing CMR for other clinical reasons not influencing cardiac function (control group)
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2009-06-16 (Actual); Primary Completion 2009-11-24 (Actual); Study Completion 2009-11-24 (Actual)

PRIMARY OUTCOMES:
Right and left atrial volume | Day of CMR (baseline only, no intervention)
  Measurement of maximal volume (at end of systole), volume before atrial contraction (in late diastole), and minimal volume (at end of diastole) of both atria.

SECONDARY OUTCOMES:
Blood flow across the atrio-ventricular valves | Day of CMR (baseline only, no intervention)
  Phase contrast measurement of blood flow across the atrio-ventricular and the ventriculo-arterial valves, respectively, to serve as an internal validation of total atrial emptying volumes, as well as to contribute maximum early and late diastolic velocities.

CONTACTS AND LOCATIONS:
Overall Officials: Emanuela R Valsangiacomo Buechel, Prof., Principal Investigator — University Children's Hospital Zürich, Switzerland
Locations (1):
- University Children's Hospital Zürich, Switzerland, Zurich, Canton of Zurich, Switzerland